CLINICAL TRIAL: NCT06064422
Title: Adaptation of a Behavioral Activation Treatment to Treat Depression in Autistic Adults
Brief Title: Adapting BA for Minimally Verbal Autistic Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Vanessa H. Bal, PhD, Associate Professor; Karmazin & Lillard Chair in Adult Autism, Rutgers, The State University of New Jersey, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro 2021001254
Record Dates: First submitted 2023-09-25; First posted 2023-10-03 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Autism; Depression; Autism Spectrum Disorder With Impaired Functional Language; Autism Spectrum Disorder
Keywords: behavioral activation
MeSH Terms: conditions — Autistic Disorder; Depression; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BeatIt-MV Treatment Group (Experimental): Participants, along with support persons, will complete 12 weekly sessions of the BeatIt-MV intervention. The support person will complete an initial session before commencement of the 12 weekly sessions.
  Interventions: Behavioral: BeatIt-MV

INTERVENTIONS:
Behavioral: BeatIt-MV — BeatIt-MV, designed to be implemented with minimally verbal autistic individuals, is an adaptation of BeatIt-2. The intervention aims to improve mood and decrease depressive symptoms through an increase in meaningful engagement in recreational, domestic, and social/leisure activities.

SUMMARY:
The present study aims to adapt and evaluate the feasibility of the BeatIt-2 behavioral activation intervention for people with intellectual disabilities and low mood to be implemented with minimally verbal autistic individuals.

DETAILED DESCRIPTION:
Aim 1. The first phase of the project will focus on adapting the BeatIt-2 manual to consider specific needs of MV autistic adults. This procedure includes an intervention development group (IDG), for which MV autistic adults and their supporters (i.e., someone identified as a source of support they can work with) will be recruited. Aim 2. During the following phase of the project, a feasibility trial will be conducted. Using the treatment manual and study procedures adapted and refined in phase 1, the trial will examine the feasibility and acceptability of BeatIt-MV.

ELIGIBILITY:
Inclusion Criteria:

* Minimally verbal
* Aged 18 years or older
* Diagnosis of Autism Spectrum Disorder and clinically significant depression based on clinical best estimate diagnosis using DSM-5 or Diagnostic Manual - Intellectual Disability criteria
* Have a support person willing to participate
* Live in New Jersey or New York, or be within travel distance to Rutgers University

Exclusion Criteria:

* Not able to engage in treatment in English
* current engagement in other treatment for depression
* conditions that may preclude engagement in treatment sessions (e.g., active psychosis, unmanaged seizures)
* high suicide risk (i.e., with a clear plan, expressed intent or recent documented attempts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Glasgow Depression Scale for Intellectual Disability (GDS) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The GDS is a 20-item self- and caregiver-reported questionnaire of psychological function over the past week with all items on a "0" (Never/No) to 2 (Always/A lot) scale. Higher scores equal more distress. Scores range from 0-32. The expected change is a decrease in the score.
Anxiety Depression and Mood Scale (ADAMS) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The ADAMS is a 20-item caregiver-reported questionnaire of psychological function over the past week with all items on a "0" (Never/No) to 2 (Always/A lot) scale. Higher scores equal more distress. Total scores range from 0-84. The expected change is a decrease in the score.
Mood, Interest, & Pleasure Questionnaire (MIPQ) | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The MIPQ is a 25-item caregiver-reported questionnaire of behaviors over the past week with all items on a "0" (Never) to 4 (All the time) scale. Higher scores equal more distress. Total scores range from 0-100. The expected change is a decrease in the score.

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scale, 3rd edition (VABS-3) | Week 1 (initial assessment) to week 22 (follow-up)
  The VABS-3 is a 381-item caregiver-reported measure of adaptive behavior. All items in the measure ask the frequency at which the participants performs a behavior, from 0 (never) to 2 (usually). Scores are age-referenced standard scores. Domain scores range from 20-140. Lower scores indicate more lower adaptive behavior. The expected change is an increase in the score.
Shalock Quality of Life Questionnaire | Week 1 (initial assessment) to week 16 (outcome) to week 22 (follow-up)
  The Shalock Quality of Life Questionnaire is a 40-item self- and caregiver-reported measure of quality of life. Each question prompts the informant to choose one of three options (differing by item) based on which seems most appropriate to them. Higher scores indicate lower quality of life. Domain scores range from 10-30. The expected change is a decrease in score.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Bal, PhD, Principal Investigator — Rutgers University - New Brunswick
Locations (1):
- Rutgers University - New Brunswick, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT06064422/ICF_000.pdf